CLINICAL TRIAL: NCT05592756
Title: Secondary Attack Rate Measles Vaccine In Second Situation Contacts Cases Confirmed
Status: Completed | Type: Observational
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 003/2019
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Measles
Keywords: soroprotegido
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be an epidemiological inquiry, in communicating confirmed measles cases. The contacts of the index cases will be asked about the measles diagnosis and previous measles vaccination, and will have their vaccination cards checked. They will also be asked about blocking vaccination (opportune or not opportune) and about the development or not of symptoms. Thus, the investigators will have a group of people exposed to infection with a history of vaccination for measles prior to the outbreak versus a group of people exposed without previous vaccination. The frequency of measles cases will be compared in those two groups, allowing to analyze the effectiveness of the vaccine for individual protection. The effectiveness of the vaccine in preventing the spread of the disease will be analyzed, comparing the relative risk of the vaccine history of contact, in the subgroups of index cases with and without previous measles vaccination.

The proposed study will involve the collection and analysis of contact data from measles cases oriented to compare vaccinated and unvaccinated, differing from health surveillance actions. This is based on an exhaustive search for contacts of measles cases, preferably aimed at detecting susceptible individuals, with the purpose of implementing blocking vaccination and interrupting the transmission chain.

The proposed study seeks a representation of contacts, without the intention of being exhaustive in the search and detection, but prioritizing selection without bias for one of the exposure groups (vaccination).

The results may provide technical and scientific support for future decisions by the Ministry of Health regarding the primary immunization schedule, the priority of the age group in vaccination campaigns, the identification of susceptible individuals, and the assessment of the need for a 3rd dose of the vaccine, for measles.

DETAILED DESCRIPTION:
This is a retrospective cohort study in which measles case contacts will be categorized according to their vaccination history and the secondary attack rate will be compared in vaccinated and non-vaccinated nodes.

ELIGIBILITY:
Inclusion Criteria:

* Characterize contact with confirmed case of measles at home, waiting room, work, etc.
* Both sexes.
* Willingness to answer the study questionnaire.
* Have had contact with the index case, 6 days before the appearance of the rash, up to 18 days after.
* Have proof of vaccination (or authorize access to health unit vaccination records) or if you no longer have a vaccination card, state whether you have had a vaccine in the past or not.
* Willingness to provide name, address, telephone and other information so that the principal investigator and his team can contact you, if necessary (example: in case of missed visit).
* Willingness to strictly follow the study protocol.
* At least one of the legal guardians for the research participants must be able to understand and sign the Free and Informed Consent Form. If those responsible are unable to sign (illiterate), the IC can be signed by an impartial witness who has accompanied the entire procedure
* For those over 6 years old, and under 18 years old, ability to understand and sign the Informed Consent Form.
* For those over 18, ability to understand and sign the Informed Consent Form.

Exclusion Criteria:

* Contact with the index case outside the contagion period, that is, after 18 days.
* Inform that you do not know the vaccination status.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Communicants referring to index cases will be interviewed. Approximately 846 contacts, with 5% of losses this amount will be 890 contacts (445 vaccinated and 445 not vaccinated). Assuming an average of 20 contacts per index case, we will need approximately 45 index cases.
Sampling Method: Non-Probability Sample
Enrollment: 2964 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Measles case after index case | 18 days after the index case
  Measles case after index case, confirmed by laboratory or epidemiological link

CONTACTS AND LOCATIONS:
Locations (1):
- Eliane Matos dos Santos, Rio de Janeiro, Brazil